CLINICAL TRIAL: NCT07189780
Title: Impact of Two Different Anterior Rectal Wall Mobilization Techniques on Postoperative Outcomes in Female Patients With Mid-low Rectal Cancer: a Multicenter, Prospective, Randomized Controlled Clinical Trial.
Brief Title: Comparison of Different Surgical Approaches in Female Rectal Cancer.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Wuhan TongJi Hospital (Other); Zhejiang Cancer Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-290
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group:Entering the dissection plane by incising the peritoneum precisely at the lowest point of the peritoneal reflection.
  Interventions: Procedure: Surgical approach
- Control Group (Active Comparator): Control Group:Entering the dissection plane by incising the peritoneum 0.5-1 cm above the lowest point of the peritoneal reflection.
  Interventions: Procedure: Surgical approach

INTERVENTIONS:
Procedure: Surgical approach — Control Group:Incising the peritoneum 0.5-1 cm above the lowest point of the peritoneal reflection to enter the dissection plane.
  Experimental Group:Incising the peritoneum precisely at the lowest point of the peritoneal reflection (in the rectovesical or rectouterine pouch) to enter the dissection plane.

SUMMARY:
Mid-to-low rectal cancer exhibits an extremely high incidence rate in China. Currently, the primary treatment approach for mid-to-low rectal cancer remains surgical intervention, with total mesorectal excision (TME) being the mainstream procedure. In male patients, Heald, Chi Pan , Wei Hongbo , and others have proposed different dissection techniques for the anterior rectal wall. Partial or complete preservation of Denonvilliers Fascia (DVF) during conventional TME (as proposed by Heald) has been shown to significantly reduce intraoperative bleeding and improve postoperative urodynamic function, urinary continence, and sexual function . However, these studies focused exclusively on male patients and did not include female subjects.

In our previous research, we proposed that females do not possess an anatomical structure equivalent to the male DVF. Furthermore, compared to entering the dissection plane by incising the peritoneum 0.5-1 cm above the lowest point of the peritoneal reflection, initiating the peritoneal incision precisely at the lowest point of the peritoneal reflection better ensures the integrity of the mesorectum and vaginal structures, reduces intraoperative bleeding, provides a more favorable operative field, and avoids damage to physiological structures while ensuring complete tumor resection, thereby promoting postoperative recovery. Thus, we concluded that this plane represents the optimal surgical dissection plane for the anterior rectal wall during TME in female patients with mid-to-low rectal cancer without anterior wall invasion.

Since our prior study combined anatomical and clinical retrospective research, we have initiated a prospective multicenter randomized controlled trial to further validate these clinical findings. This study aims to demonstrate that entering the dissection plane at the lowest point of the peritoneal reflection during mid-to-low rectal cancer surgery improves prognosis in female patients, providing high-level evidence-based medical support for the adoption of this technique and establishing the optimal surgical approach for female rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed rectal adenocarcinoma.
2. Female patients scheduled to undergo laparoscopic total mesorectal excision (TME).
3. Body mass index (BMI) ≤ 30 kg/m².
4. Tumors with the distal margin located ≤ 10 cm from the anal verge.
5. Absence of distant metastases (e.g., to the liver, lungs, or other organs).

Exclusion Criteria:

1. Presence of severe pre-existing comorbidities (e.g., significant hepatic, renal, cardiac, pulmonary, or coagulation dysfunction).
2. History of malignancy in other organs.
3. Patients requiring emergency surgery due to conditions such as acute perforation or obstruction.
4. Intraoperative findings of tumor invasion into adjacent organs necessitating multivisceral resection or palliative resection.
5. Previous history of anorectal or rectal surgery. 6Preoperative magnetic resonance imaging (MRI) indicating invasion of the anterior rectal wall.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Estimated Blood Loss | 2-6hours

IPD SHARING:
Plan to Share IPD: Yes